CLINICAL TRIAL: NCT07104786
Title: Effectiveness of Obeticholic Acid Versus Vitamin E in Patients of Non-alcoholic Fatty Liver Disease
Brief Title: Comparison of Effectiveness of Obeticholic Acid With Vitamin E in Patients of Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Tazeen Nazar, Associate Professor of Medicine, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: No.166/RC/KEMU Date 08/06/2023
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: Obeticholic acid; Vitamin E; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — obeticholic acid; Vitamin E; Tocopherols

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial. Patients were randomly divided into two groups. Group A received 10mg Obeticholic acid once daily, whereas Group B received 400mg Vitamin E twice daily. Both groups were treated for 6 months. Changes in grade of NAFLD on ultrasound and ALT levels were monitored.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obeticholic acid (OCA) 10mg, Group A (Experimental): 45 patients received 10mg of Obeticholic acid daily for 6 months
  Interventions: Drug: Obeticholic Acid 10 MG
- Vitamin E 400mg twice daily, Group B (Active Comparator): 45 patients received 400mg of Vitamin E twice daily for 6 months
  Interventions: Dietary Supplement: Vitamin E 400mg

INTERVENTIONS:
Drug: Obeticholic Acid 10 MG — 10mg OCA was given once daily for 6 months
  Other Names: OCA
  Arms: Obeticholic acid (OCA) 10mg, Group A
Dietary Supplement: Vitamin E 400mg — Vitamin E 400mg was given twice daily for 6 months
  Other Names: Evion
  Arms: Vitamin E 400mg twice daily, Group B

SUMMARY:
This study was conducted on patients presenting to Mayo Hospital, Lahore from 24th August, 2023 till 23rd May, 2024. Ninety patients conforming to the inclusion criteria were selected via simple random sampling technique and divided into two groups. Group A received Obeticholic acid 10mg once a day and Group B received Vitamin E 400mg twice a day. Both treatments were given for 6 months alongwith clear written and informed instructions regarding lifestyle modification. Patients were followed at 3 and 6 months with ultrasound abdomen and serum alanine transferase levels.

DETAILED DESCRIPTION:
This study was conducted in the Liver Clinic, patients presenting to the out-patients department and admitted on the Medical floor of Mayo Hospital, Lahore after taking approval from the Institutional Review Board of King Edward Medical University (KEMU) No. 166/RC/KEMU, dated 08-06-2023. A sample size of 90 patients (45 patients in each group) was estimated using 5% level of significance, 90% power of test with expected percentage improvement of fibrosis by ≥ 1 grade in obeticholic acid 10mg as 21% and vitamin E as 50%. Simple random sampling technique was employed in patient selection. Consenting adults of either gender between 18-75 years of age, diagnosed to have any grade of NAFLD on ultrasonography (Grade 1 to 3) and raised ALT >1.5 times the upper normal limit. (Normal reference <40 IU in males, <32 IU females) were included in the study. Patients with significant alcohol intake (more than 20 g/day in women and >30g/day in men), history of taking drugs that may cause fatty liver (i.e. tamoxifen, valproic acid, amiodarone, methotrexate, steroid, oral contraceptive pills), patients with co-morbid conditions like Diabetes, Chronic Obstructive Pulmonary Disease, Chronic Kidney Disease, Congestive Cardiac Failure, Hypothyroidism were excluded from the study. Pregnant and lactating females, patients with history of recent myocardial infarction, cirrhosis (decompensated liver) and portal hypertension, patients taking drugs known to have significant interaction with Obeticholic acid or vitamin E including cholestyramine, theophylline and colestipol were also excluded from the study protocol. After taking informed written and verbal consent, all patients conforming to the selection criteria were enrolled in the study. The patients were randomly enrolled into two groups of 45 patients each, by computer generated lottery method. Demographic details along with initial investigations were obtained i.e., liver function test (ALT) and Ultrasound Abdomen.

Group A patients were treated with Obeticholic acid 10mg once a day whereas Group B patients were treated with Vitamin E 400mg twice a day. Total duration of treatment was 6 months. Both groups of patients were advised dietary and lifestyle modification through a separate handout and counselling session. The patients were followed up at 3 and 6 months, at 3 months to ensure compliance to lifestyle and dietary modifications and medication, also ALT levels were checked.

At 6 months follow-up, patients were subjected to ultrasound evaluation as well as ALT level measurement. Data was recorded on a predesigned proforma. Effectiveness was defined in terms of improvement on ultrasonography by at least one grade or reduction of ALT by at least 25% from the baseline or both. All patients were guided to report if they experienced any adverse effects of medications. Non-compliance to medication due to any cause resulted in exclusion from the study.

Data was entered and analyzed using computer software SPSS 26.0 version. Quantitative variables like age, weight, ALT levels were presented as mean ± SD. Qualitative variables like gender, grade of NAFLD were presented as frequency and percentage. Independent sample t test was used to compare pre and post treatment ALT levels in both the groups. Chi square was applied for comparison of NAFLD grading pre and post treatment in both groups. p-value ≤0.05 was taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults of either gender between 18-75 years of age
* Any grade of NAFLD on ultrasonography (Grade 1 to 3)
* Raised ALT >1.5 times the upper normal limit. (Normal reference <40 IU in males, <32 IU females)

Exclusion Criteria:

* Patients with significant alcohol intake (more than 20 g/day in women and >30g/day in men)
* History of taking drugs that may cause fatty liver (i.e. tamoxifen, valproic acid, amiodarone, methotrexate, steroid, oral contraceptive pills)
* Patients with co-morbid conditions like Diabetes, Chronic Obstructive Pulmonary Disease, Chronic Kidney Disease, Congestive Cardiac Failure, Hypothyroidism
* Pregnant and lactating females
* Patients with history of recent myocardial infarction, cirrhosis (decompensated liver) and portal hypertension
* Patients taking drugs known to have significant interaction with Obeticholic acid or vitamin E including cholestyramine, theophylline and colestipol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Change in grade of NAFLD on ultrasound | 6 months
  Improvement/ reduction on ultrasonography of at least one grade of NAFLD from baseline
Reduction of ALT levels | 6 months
  25% reduction of ALT levels from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tazeen Nazar, MBBS,FCPSMed, Study Director — King Edward Medical University
Locations (1):
- King Edward Medical University, Mayo Hospital, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
To maintain confidentiality.

REFERENCES:
- [Background] Rinella ME, Lominadze Z, Loomba R, Charlton M, Neuschwander-Tetri BA, Caldwell SH, Kowdley K, Harrison SA. Practice patterns in NAFLD and NASH: real life differs from published guidelines. Therap Adv Gastroenterol. 2016 Jan;9(1):4-12. doi: 10.1177/1756283X15611581. PMID 26770262
- [Background] El Hadi H, Vettor R, Rossato M. Vitamin E as a Treatment for Nonalcoholic Fatty Liver Disease: Reality or Myth? Antioxidants (Basel). 2018 Jan 16;7(1):12. doi: 10.3390/antiox7010012. PMID 29337849
- [Background] Zhou J, Zhou F, Wang W, Zhang XJ, Ji YX, Zhang P, She ZG, Zhu L, Cai J, Li H. Epidemiological Features of NAFLD From 1999 to 2018 in China. Hepatology. 2020 May;71(5):1851-1864. doi: 10.1002/hep.31150. PMID 32012320
- [Background] Roy PP, Mahtab MA, Rahim MA, Yesmin SS, Islam SB, Akbar SMF. Treatment of Nonalcoholic Steatohepatitis by Obeticholic Acid: Current Status. Euroasian J Hepatogastroenterol. 2022 Jul;12(Suppl 1):S46-S50. doi: 10.5005/jp-journals-10018-1360. PMID 36466097
- [Background] Kamrul-Hasan A, Mondal S, Nagendra L, Sasikanth T, Ahammed A, Rahman S, Wickramarachchi A, Parajuli N, Khatiwada S, Dutta D. Role of Obeticholic Acid, a Farnesoid X Receptor Agonist, in Nonalcoholic Fatty Liver Disease: A Systematic Review and Meta-analysis. touchREV Endocrinol. 2024 Oct;20(2):54-61. doi: 10.17925/EE.2024.20.2.8. Epub 2024 Oct 9. PMID 39526049
- [Background] 23. Abo Farrag GA, Afifi MA, El-Aziz SA, Ghoname MM, Ali AA. Role of Farnesoid X Receptor Ligand Obeticholic Acid Versus Vitamin E for Patients with Nonalcoholic Steatohepatitis. Al-Azhar International Medical Journal 2024; 5(10), Article 25. DOI: https://doi.org/10.58675/2682-339X.2706
- [Background] Karedath J, Javed H, Ahsan Talpur F, Lal B, Kumari A, Kivan H, Anirudh Chunchu V, Hirani S. Effect of Vitamin E on Clinical Outcomes in Patients With Non-alcoholic Fatty Liver Disease: A Meta-Analysis. Cureus. 2022 Dec 21;14(12):e32764. doi: 10.7759/cureus.32764. eCollection 2022 Dec. PMID 36686141
- [Background] Zhao J, Li B, Zhang K, Zhu Z. The effect and safety of obeticholic acid for patients with nonalcoholic steatohepatitis: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2024 Feb 16;103(7):e37271. doi: 10.1097/MD.0000000000037271. PMID 38363900
- [Background] 20. Aishwarya TS, Mounika N, Vishwakarma G, Adela R, Effect of obeticholic acid in non-alcoholic fatty liver disease (NAFLD) and non-alcoholic steatohepatitis (NASH) patients: a systematic review and meta-analysis, RPS Pharmacy and Pharmacology Reports, Volume 1, Issue 1, September 2022, rqac001, https://doi.org/10.1093/rpsppr/rqac001
- [Background] Paternostro R, Trauner M. Current treatment of non-alcoholic fatty liver disease. J Intern Med. 2022 Aug;292(2):190-204. doi: 10.1111/joim.13531. Epub 2022 Jul 7. PMID 35796150
- [Background] Kulkarni AV, Tevethia HV, Arab JP, Candia R, Premkumar M, Kumar P, Sharma M, Reddy DN, Padaki NR. Efficacy and safety of obeticholic acid in liver disease-A systematic review and meta-analysis. Clin Res Hepatol Gastroenterol. 2021 May;45(3):101675. doi: 10.1016/j.clinre.2021.101675. Epub 2021 Mar 17. PMID 33722778
- [Background] Li J, Zou B, Yeo YH, Feng Y, Xie X, Lee DH, Fujii H, Wu Y, Kam LY, Ji F, Li X, Chien N, Wei M, Ogawa E, Zhao C, Wu X, Stave CD, Henry L, Barnett S, Takahashi H, Furusyo N, Eguchi Y, Hsu YC, Lee TY, Ren W, Qin C, Jun DW, Toyoda H, Wong VW, Cheung R, Zhu Q, Nguyen MH. Prevalence, incidence, and outcome of non-alcoholic fatty liver disease in Asia, 1999-2019: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2019 May;4(5):389-398. doi: 10.1016/S2468-1253(19)30039-1. Epub 2019 Mar 20. PMID 30902670
- [Background] Riazi K, Azhari H, Charette JH, Underwood FE, King JA, Afshar EE, Swain MG, Congly SE, Kaplan GG, Shaheen AA. The prevalence and incidence of NAFLD worldwide: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2022 Sep;7(9):851-861. doi: 10.1016/S2468-1253(22)00165-0. Epub 2022 Jul 5. PMID 35798021
- [Background] Le MH, Yeo YH, Li X, Li J, Zou B, Wu Y, Ye Q, Huang DQ, Zhao C, Zhang J, Liu C, Chang N, Xing F, Yan S, Wan ZH, Tang NSY, Mayumi M, Liu X, Liu C, Rui F, Yang H, Yang Y, Jin R, Le RHX, Xu Y, Le DM, Barnett S, Stave CD, Cheung R, Zhu Q, Nguyen MH. 2019 Global NAFLD Prevalence: A Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2022 Dec;20(12):2809-2817.e28. doi: 10.1016/j.cgh.2021.12.002. Epub 2021 Dec 7. PMID 34890795
- [Background] Bril F, Biernacki DM, Kalavalapalli S, Lomonaco R, Subbarayan SK, Lai J, Tio F, Suman A, Orsak BK, Hecht J, Cusi K. Role of Vitamin E for Nonalcoholic Steatohepatitis in Patients With Type 2 Diabetes: A Randomized Controlled Trial. Diabetes Care. 2019 Aug;42(8):1481-1488. doi: 10.2337/dc19-0167. Epub 2019 May 21. PMID 31332029
- [Background] Hindson J. Obeticholic acid for the treatment of NASH. Nat Rev Gastroenterol Hepatol. 2020 Feb;17(2):66. doi: 10.1038/s41575-020-0264-1. No abstract available. PMID 31919473
- [Background] Amanullah I, Khan YH, Anwar I, Gulzar A, Mallhi TH, Raja AA. Effect of vitamin E in non-alcoholic fatty liver disease: a systematic review and meta-analysis of randomised controlled trials. Postgrad Med J. 2019 Nov;95(1129):601-611. doi: 10.1136/postgradmedj-2018-136364. Epub 2019 Aug 21. PMID 31434683
- [Background] Perumpail BJ, Li AA, John N, Sallam S, Shah ND, Kwong W, Cholankeril G, Kim D, Ahmed A. The Role of Vitamin E in the Treatment of NAFLD. Diseases. 2018 Sep 24;6(4):86. doi: 10.3390/diseases6040086. PMID 30249972
- [Background] Younossi ZM, Ratziu V, Loomba R, Rinella M, Anstee QM, Goodman Z, Bedossa P, Geier A, Beckebaum S, Newsome PN, Sheridan D, Sheikh MY, Trotter J, Knapple W, Lawitz E, Abdelmalek MF, Kowdley KV, Montano-Loza AJ, Boursier J, Mathurin P, Bugianesi E, Mazzella G, Olveira A, Cortez-Pinto H, Graupera I, Orr D, Gluud LL, Dufour JF, Shapiro D, Campagna J, Zaru L, MacConell L, Shringarpure R, Harrison S, Sanyal AJ; REGENERATE Study Investigators. Obeticholic acid for the treatment of non-alcoholic steatohepatitis: interim analysis from a multicentre, randomised, placebo-controlled phase 3 trial. Lancet. 2019 Dec 14;394(10215):2184-2196. doi: 10.1016/S0140-6736(19)33041-7. Epub 2019 Dec 5. PMID 31813633
- [Background] Zhang DY, Zhu L, Liu HN, Tseng YJ, Weng SQ, Liu TT, Dong L, Shen XZ. The protective effect and mechanism of the FXR agonist obeticholic acid via targeting gut microbiota in non-alcoholic fatty liver disease. Drug Des Devel Ther. 2019 Jul 5;13:2249-2270. doi: 10.2147/DDDT.S207277. eCollection 2019. PMID 31308634
- [Background] Neuschwander-Tetri BA, Loomba R, Sanyal AJ, Lavine JE, Van Natta ML, Abdelmalek MF, Chalasani N, Dasarathy S, Diehl AM, Hameed B, Kowdley KV, McCullough A, Terrault N, Clark JM, Tonascia J, Brunt EM, Kleiner DE, Doo E; NASH Clinical Research Network. Farnesoid X nuclear receptor ligand obeticholic acid for non-cirrhotic, non-alcoholic steatohepatitis (FLINT): a multicentre, randomised, placebo-controlled trial. Lancet. 2015 Mar 14;385(9972):956-65. doi: 10.1016/S0140-6736(14)61933-4. Epub 2014 Nov 7. PMID 25468160
- [Background] Attia SL, Softic S, Mouzaki M. Evolving Role for Pharmacotherapy in NAFLD/NASH. Clin Transl Sci. 2021 Jan;14(1):11-19. doi: 10.1111/cts.12839. Epub 2020 Aug 25. PMID 32583961
- [Background] Mundi MS, Velapati S, Patel J, Kellogg TA, Abu Dayyeh BK, Hurt RT. Evolution of NAFLD and Its Management. Nutr Clin Pract. 2020 Feb;35(1):72-84. doi: 10.1002/ncp.10449. Epub 2019 Dec 16. PMID 31840865
- [Background] Huang DQ, Singal AG, Kono Y, Tan DJH, El-Serag HB, Loomba R. Changing global epidemiology of liver cancer from 2010 to 2019: NASH is the fastest growing cause of liver cancer. Cell Metab. 2022 Jul 5;34(7):969-977.e2. doi: 10.1016/j.cmet.2022.05.003. Epub 2022 Jun 3. PMID 35793659
- [Background] Tan DJH, Setiawan VW, Ng CH, Lim WH, Muthiah MD, Tan EX, Dan YY, Roberts LR, Loomba R, Huang DQ. Global burden of liver cancer in males and females: Changing etiological basis and the growing contribution of NASH. Hepatology. 2023 Apr 1;77(4):1150-1163. doi: 10.1002/hep.32758. Epub 2022 Sep 12. PMID 36037274